CLINICAL TRIAL: NCT07404514
Title: Prospective and Retrospective Observational Study on Longitudinal Ulnar Deficit: Analysis of Existing Medical Data and Parental Questionnaires
Brief Title: Longitudinal Ulnar Deficiency: Analysis of Existing Medical Data and Parental Questionnaires
Acronym: ULNEER
Status: Not yet recruiting | Type: Observational
Sponsor: Hopitaux de Saint-Maurice (Other)
Responsible Party: Sponsor
Other Study IDs: ULNEER; 2025-A02482-47 (Other: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2026-02-02; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Ulnar Hand Deformity; Ulnar Longitudinal Deficit; Occupational Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ulnar Longitudinal Deficiency Observational Cohort: This arm represents a non-interventional observational cohort of children and adolescents with ulnar longitudinal deficiency.
  No intervention is assigned as part of the study. Clinical, radiological, and rehabilitation data are collected retrospectively from existing medical records and prospectively through parent-reported outcome questionnaires (PROMIS and ABILHAND-Kids-CP), without any modification of standard clinical care.

SUMMARY:
The management of patients with longitudinal ulnar deficiency is a clinical challenge due to the rarity of this condition and the wide variety of its manifestations. In particular, there is no consensus in the literature on the indications for surgery.

The aim of this research is to improve understanding and management of this malformation by analyzing existing data from patient medical follow-up.

No new clinical evaluations or occupational therapy assessments will be performed specifically for this study.

The analysis will be based on previous medical and paramedical data (consultation reports, imaging, occupational therapy assessments, etc.) in order to better describe the functional evolution of patients and identify the decision-making criteria that guide surgical management.

Parents will also receive standardized questionnaires (PROMIS and ABILHAND-Kids-CP) to gather their perceptions of their child's quality of life and independence.

The results will be used to propose recommendations for a more consistent and multidisciplinary assessment of longitudinal ulnar deficit in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral or bilateral ulnar hand deformity, whether operated on or not
* Follow-up at CEREFAM and/or Trousseau Hospital
* Complete medical records containing previous assessments

Exclusion Criteria:

* Non-French-speaking patient
* No preoperative or postoperative assessment

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of children and adolescents aged 3 to 18 years diagnosed with ulnar longitudinal deficiency, either unilateral or bilateral.
  Participants are followed at a tertiary referral center for upper limb malformations and have available medical records allowing retrospective data extraction. Parent-reported outcome measures are collected prospectively as part of the study without modifying standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Upper limb function and health-related quality of life (PROMIS Upper Extremity and ABILHAND-Kids) | From baseline to study completion (up to 10 months)
  Upper limb function and health-related quality of life will be assessed using validated parent-reported outcome measures, including the Pediatric Outcomes Measurement Information System (PROMIS) Upper Extremity Pediatric questionnaire and the ABILHAND-Kids questionnaire.
  PROMIS Upper Extremity Pediatric questionnaire scores range from 0 to 100, with higher scores indicating better upper limb function and health-related quality of life.
  ABILHAND-Kids scores range from 0 to 100, with higher scores indicating better manual ability.

SECONDARY OUTCOMES:
Upper limb functional ability score | From baseline to study completion (up to 10 months)
  Upper limb functional ability will be assessed using the ABILHAND-Kids questionnaire (Assessment of Manual Ability for Children).
  The ABILHAND-Kids score ranges from 0 to 100, with higher scores indicating better manual ability.
Pediatric upper limb function | From baseline to study completion (up to 10 months)
  Upper limb function will be assessed using the Pediatric Outcomes Measurement Information System (PROMIS) Upper Extremity Pediatric questionnaire.
  Scores range from 0 to 100, with higher scores indicating better upper limb function.
Pediatric health-related quality of life | From baseline to study completion (up to 10 months)
  Health-related quality of life assessed using the PROMIS pediatric quality of life questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Paris Est Val-de-Marne - Centre de Référence des Malformations des Membres, Saint-Maurice, France

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the small sample size, the pediatric population involved, and the need to ensure participant confidentiality in accordance with applicable data protection regulations.